CLINICAL TRIAL: NCT06048757
Title: Effectiveness of the Mobile Application-delivered Resistance Program for Children and Adolescents With Type 1 Diabetes (Diactive-1) on Insulin Requirements: Protocol for a Randomized Controlled Trial
Brief Title: Mobile Application-delivered Resistance Program for Children and Adolescents With Type 1 Diabetes (Diactive-1)
Acronym: Diactive-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Miguel Servet (Other)
Collaborators: Complejo Hospitalario de Navarra (Other); Universidad Pública de Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGH_Diactive1_2023
Record Dates: First submitted 2023-08-28; First posted 2023-09-21 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Type 1 Diabetes
Keywords: mHealth; Resistance exercise; Insulin sensitivity; Glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental app intervention group (Experimental): The intervention in the experimental group will center around the use of a mobile application (i.e., device), namely the Diactive-1 app.
  Interventions: Device: Diactive-1 application
- Waiting-list control group (No Intervention): This arm will not complete an intervention. Participants will be instructed to continue to follow their normal daily diabetes care plan (i.e., standard care). This group will be granted access to the app following the intervention.

INTERVENTIONS:
Device: Diactive-1 application — Participants will engage in 24 weeks resistance exercise program with goal of maintaining at least 3 sessions per week with 4-5 exercises per session (13-33 minutes). The training intervention will comprise 3-4 sets of 6-12 repetitions and will consist of a combination of exercises for the upper and lower body and the core, utilizing the participants' body weight as the primary resistance or auxiliary materials such as elastic bands and a water-fillable kettlebell. The load and intensity of the exercise will be based on the number of repetitions, the resistance of the elastic bands and/or the weight of the aquaball, as well as the difficulty of the exercises. A mobile application known as Diactive-1 will be utilized.
  Arms: Experimental app intervention group

SUMMARY:
This project involves a two-arm randomized controlled trial (RCT) designed to assess the feasibility, acceptability, and preliminary efficacy of a mobile application aimed at prescribing resistance training for children and adolescents with type 1 diabetes (Diactive-1). The program will span 24 weeks, with a minimum weekly frequency of 3 sessions. The researchers aim to recruit 52 participants but will enroll additional participants to account for potential withdrawals and ensure compliance with the desired sample size. The primary objective of the study is to evaluate the impact of the Diactive-1 mobile application on insulin requirements in children and adolescents with Type 1 Diabetes. Additionally, the researchers will investigate the effects of the Diactive-1 program on secondary parameters such as glycemic control, cardiometabolic indicators, physical fitness, and daily physical activity, among others. The hypothesis posits that personalized training through a mobile application, primarily focusing on muscular strength, will effectively reduce the daily insulin dosage in children and adolescents with type 1 diabetes.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the effectiveness of the Diactive-1 mobile application, which offers personalized resistance training, in reducing daily insulin requirements among children and adolescents with type 1 diabetes.

To achieve this objective, researchers will conduct a 24 weeks randomized controlled trial involving at least 52 participants diagnosed with type 1 diabetes. The study will consist of two groups: an experimental group utilizing the Diactive-1 application and a control group receiving standard treatment. Participant allocation to either group will be determined through central randomization.

The Diactive-1 intervention encompasses several key features, including: (i) tailoring exercises based on initial physical fitness levels; (ii) adjusting the previous exercise to the glucose level measured through an interstitial glucose monitor or entered manually before the training session; (iii) monitoring heart rate during exercise; (iv) providing the flexibility to train with or without equipment, individually or with a partner; (v) dispensing diabetes management advice before and after each training session; and (vi) adapting training progressions based on session adherence. A face-to-face session will be conducted before commencing the intervention to ensure that participants are familiar with the fundamental movements, thus reducing the risk of potential muscle injuries.

ELIGIBILITY:
Inclusion Criteria:

* Aged 8-18 years old
* At least 6 months post-diagnosis for type 1 diabetes
* Ability to complete measures and intervention program in Spanish
* Access to broadband or cellular internet
* Patients who signed the informed consent form prior to participation; for minors, a legal representative must provide consent and sign the informed consent form.

Exclusion Criteria:

* Any comorbidity limiting the capacity to participate in physical activity or inadequate understanding of the Spanish language.
* Participants will be excluded if they don't have access to the internet, lack a smartphone or tablet, or are unable to use the application.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2023-08-20 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Change in daily insulin dose requirement | Baseline, 12 and 24 weeks
  The daily insulin dose requirements will be measured in units per kilogram of body weight. Assessment will rely on participant-reported data from insulin pumps or injection logs, gathered for 9 days prior to the intervention, at 12 weeks, and after the intervention.

SECONDARY OUTCOMES:
Change in glycated hemoglobin | Baseline and 24 weeks
  Glycated hemoglobin (measured in percent)
Number of participants with good glycemic control | Baseline and 24 weeks
  Number of participants with a glycated hemoglobin level lower than 7%
Change in time in range | Baseline and 24 weeks
  The percentage of time a person spends with their blood glucose levels in the target range (70-180 mg/dL or 3.9-10 mmol/L) (measured in percent)
Change in time below range | Baseline and 24 weeks
  The percentage of time a person spends with their blood glucose levels below the target range (<70 mg/dL or <3.9 mmol/L, i.e., hypoglycemia) (measured in percent)
Change in time above range | Baseline and 24 weeks
  The percentage of time a person spends with their blood glucose levels above the target range (>180 mg/dL or 10 mmol/L, i.e., hyperglycemia) (measured in percent).
Change in glycemic variability | Baseline and 24 weeks
  Glycemic variability measures the fluctuation in blood glucose levels over time, expressed as a percentage. Lower glycemic variability indicates more stable levels, while higher glycemic variability suggests greater fluctuations.
Change in compliance with 24-hour movement behaviors | Baseline and 24 weeks
  Physical activity at different intensities (average min/day), sedentary time (average min/day) and sleep (average min/day) will be measured using GENEActive accelerometers and self-reported questionnaires
Change in physical activity | Baseline, 12 and 24 weeks
  Physical activity will be estimated using the GENEActive triaxial accelerometer (ActivInsights) and measured in minutes per day
Change in self-reported physical activity | Baseline and 24 weeks
  Aerobic and muscle-strengthening activities will be assessed using two separate ad hoc questions. Participants will have response options ranging from 0 to 7 days per week, with increments of 1 day
Change in sedentary behaviors | Baseline and 24 weeks
  Sedentary behaviors will be self-reported using the Youth Leisure-Time Sedentary Behavior Questionnaire. Total daily sedentary screen time will be calculated by summing the durations of daily screen time activities. Furthermore, total screen time for both weekdays and weekends will be calculated in minutes per day
Change in sleep duration | Baseline and 24 weeks
  Sleep duration will be determined by recording the number of hours slept each day in a 9-day diary
Change in sleep quality | Baseline and 24 weeks
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index questionnaire, which evaluates seven established aspects of sleep quality: subjective sleep quality, time taken to fall asleep, duration of sleep, sleep efficiency, sleep disturbances (such as nightmares, pain, or feeling too hot or cold), use of sleep medication, and daytime dysfunction. Each question is scored on a scale from 0 to 3, with higher scores indicating more pronounced sleep disturbances.
Change in blood pressure | Baseline and 24 weeks
  Systolic and diastolic blood pressure will be measured in mmHg using a blood pressure monitor
Change in cardio-ankle vascular index (CAVI) | Baseline and 24 weeks
  Measuring Cardio-Ankle Vascular Index (measured in percent) by VaSera VS 2000 (Fukuda Denshi, Japan)
Change in pulse wave velocity | Baseline and 24 weeks
  Measuring pulse wave velocity (m/seg) by VaSera VS 2000 (Fukuda Denshi, Japan)
Change in heart rate variability | Baseline and 24 weeks
  The heart rate will be recorded by a heart rate monitor in a beat-by-beat basis.
Change in disordered eating | Baseline and 24 weeks
  Disordered eating will be screened using the mSCOFF questionnaire. This questionnaire consists of six straightforward yes/no questions. A positive response to two or more of these questions suggests a potential eating disorder, often requiring further evaluation.
Change in Health-Related Quality of Life in the context of a chronic illness | Baseline and 24 weeks
  Health-Related Quality of Life in the context of a chronic illness will be evaluated using the Spanish version of the 'Questionnaire for Young People with Diabetes' (DISABKIDS). This questionnaire consists of 12 questions about how a patient has felt in the last four weeks, with responses rated on a 5-point Likert scale from 1 (Never) to 5 (Always)
Change in Health-Related Quality of Life | Baseline and 24 weeks
  Health-Related Quality of Life will be evaluated using the Screening for and Promotion of Health-Related Quality of Life in Children and Adolescents (KIDSCREEN-10). This is a generic 10-item unidimensional instrument that assesses the functional, mental, and social aspects of well-being in children and adolescents. Each item will offer five response categories, ranging from 'never' to 'always' or from 'not at all' to 'extremely'
Change in subjective well-being | Baseline and 24 weeks
  Subjective well-being will be assessed using the 'Cuestionario Unico de Bienestar Escolar' (CUBE), which comprises five items evaluating different aspects of life satisfaction. All variables will be measured on a 10-point Likert scale ranging from 0 to 10 (0 = totally disagree, 10 = totally agree).
Change in cardiorespiratory fitness | Baseline and 24 weeks
  Measured with an incremental VO2 protocol on exercise bike by COSMED Quark CPET plus OMNIA (COSMED®, Rome, Italy) (measured in mL/kg/min and Metabolic Equivalents [METs])
Change in isometric strength | Baseline, 12 and 24 weeks
  Handgrip strength measured in kilograms using the Takei III Smedley Type Digital Dynamometer
Change in lower limb muscle dynamic strength | Baseline and 24 weeks
  Lower limb muscle strength (legs and hips) measured in kg using eGym® machines (GmbH in Munich, Germany)
Change in upper limb muscle dynamic strength | Baseline and 24 weeks
  Upper limb muscle strength (chest and arms) measured in kg using eGym® machines (GmbH in Munich, Germany)
Change in lower limb muscle power strength | Baseline and 24 weeks
  Lower limb muscle power (legs and hips) measured in watts using eGym® machines (GmbH in Munich, Germany)
Change in upper limb muscle power strength | Baseline and 24 weeks
  Upper limb muscle power (chest and arms) measured in watts using eGym® machines (GmbH in Munich, Germany)
Change in self-reported physical fitness | Baseline and 24 weeks
  The International Fitness Scale (IFIS) will be used to assess self-reported physical fitness. This scale includes five elements that will employ a 5-point Likert scale to inquire about children's overall perception of their physical fitness, as well as their perception of their cardiorespiratory fitness, muscular fitness, speed-agility, and flexibility compared to their peers. The Likert scale will provide choices ranging from 'very poor' to 'poor,' 'average,' 'good,' and 'very good' physical fitness.
Adherence to the Mediterranean Diet | Baseline and 24 weeks
  For assessing adherence to the Mediterranean Diet, the KIDMED index will be employed. This index provides a score on a scale of 0 to 12, with higher scores indicating stronger adherence.
Change in dietary behavior | Baseline and 24 weeks
  Self-reported food intake will be assessed using a food-frequency questionnaire (FFQ). The daily consumption of food and beverages will be categorized into 12 groups: dairy, meat, fish, eggs, vegetables, fruit, starch, legumes, nuts, sweets, soft drinks, and alcoholic drinks.
Change in body mass index | Baseline, 12 and 24 weeks
  Weight and height will be combined to report body mass index in kg/m^2
Change in fat mass (percentage) | Baseline, 12 and 24 weeks
  Fat mass will be measured using a dual-energy X-ray absorptiometer (DXA) and expressed as a percentage.
Change in fat mass (in kilograms) | Baseline, 12 and 24 weeks
  Fat mass will be measured using a dual-energy X-ray absorptiometer (DXA) and expressed in kilograms.
Change in lean mass | Baseline, 12 and 24 weeks
  Fat mass in kilograms will be measured using a dual-energy X-ray absorptiometer (DXA)
Change in subcutaneos adiposity | Baseline, 12 and 24 weeks
  Subcutaneos adiposity in cm^3 will be measured using a dual-energy X-ray absorptiometer (DXA)
Change in visceral adiposity | Baseline, 12 and 24 weeks
  Visceral adiposity in cm^3 will be measured using a dual-energy X-ray absorptiometer (DXA)
Change in bone mineral content | Baseline, 12 and 24 weeks
  Bone mineral content in grams will be measured using a dual-energy X-ray absorptiometer (DXA)
Change in bone mineral density | Baseline, 12 and 24 weeks
  Bone mineral density will be measured in grams/cm^2 using a dual-energy X-ray absorptiometer (DXA)
Change in blood lipids levels | Baseline and 24 weeks
  The following parameters will be evaluated: fasting total cholesterol, LDL-Cholesterol, HDL-Cholesterol, triglycerides, lipoprotein (a), and apolipoproteins A-I and B levels, measured in mg/dL.
Change in fasting glucose | Baseline and 24 weeks
  Fasting glucose will be measured in mg/dL.
Changes in liver enzymes | Baseline and 24 weeks
  The following parameters will be evaluated: alanine transaminase and aspartate aminotransferase.
Change in inadvertent hypoglycemia | Baseline and 24 weeks
  The perception of hypoglycemia will be assessed using the Clarke test, which comprises eight questions with various potential answers. A score greater than 3 indicates impaired awareness of hypoglycemia.
App usability | 24 weeks
  The usability of the app will be evaluated using the Spanish Version of the User Version of the Mobile Application Rating Scale (uMARS). This scale provides a comprehensive and objective measure of app usability and consists of 20 items. Each item is rated on a 5-point scale, ranging from 1 (inadequate) to 5 (excellent).

CONTACTS AND LOCATIONS:
Overall Officials: Antonio García-Hermoso, PhD, Principal Investigator — Fundación Miguel Servet - Navarrabiomed
Locations (2):
- Spain (2):
  - Fundación Miguel Servet/ Navarrabiomed, Pamplona, Navarre
  - Paediatric Endocrinology Unit at Hospital Universitario de Navarra, Pamplona, Navarre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hormazabal-Aguayo I, Munoz-Pardeza J, Lopez-Gil JF, Huerta-Uribe N, Chueca-Guindulain MJ, Berrade-Zubiri S, Burillo Sanchez E, Izquierdo M, Ezzatvar Y, Garcia-Hermoso A. Comprehensive management of children and adolescents with type 1 diabetes mellitus through personalized physical exercise and education using an mHealth system: The Diactive-1 study protocol. Front Endocrinol (Lausanne). 2024 Feb 6;15:1354734. doi: 10.3389/fendo.2024.1354734. eCollection 2024. PMID 38379866
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/40802196/